CLINICAL TRIAL: NCT02347761
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Efficacy and Safety Trial of 12 Weeks of Treatment With Nebulized SUN-101 in Patients With COPD: GOLDEN-3 (Glycopyrrolate for Obstructive Lung Disease Via Electronic Nebulizer)
Brief Title: Efficacy and Safety Trial of 12 Weeks of Treatment With Nebulized SUN-101 in Patients With COPD
Acronym: GOLDEN-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN101-301
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SUN-101 50 mcg BID eFlow (CS) nebulizer (Experimental): SUN-101 50 mcg twice daily (BID) eFlow (R) Closed System (CR) nebulizer
  Interventions: Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer
- SUN-101 25 mcg BID eFlow (CS) nebulizer (Experimental): SUN-101 25 mcg twice daily (BID) eFlow (R) Closed System (CR) nebulizer
  Interventions: Drug: SUN-101 25 mcg BID eFlow (CS) nebulizer
- Placebo BID eFlow (CS) nebulizer (Placebo Comparator): Placebo twice daily (BID) eFlow (R) Closed System (CR) nebulizer
  Interventions: Drug: Placebo BID eFlow Closed System (CS) nebulizer

INTERVENTIONS:
Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer — SUN-101 50 mcg twice daily (BID) eFlow Closed System (CS) nebulizer
  Arms: SUN-101 50 mcg BID eFlow (CS) nebulizer
Drug: SUN-101 25 mcg BID eFlow (CS) nebulizer — SUN-101 25 mcg twice daily (BID) eFlow Closed System (CS) nebulizer
  Arms: SUN-101 25 mcg BID eFlow (CS) nebulizer
Drug: Placebo BID eFlow Closed System (CS) nebulizer — Placebo twice daily (BID) eFlow Closed System (CS) nebulizer
  Arms: Placebo BID eFlow (CS) nebulizer

SUMMARY:
This is a trial of 12 weeks of treatment with nebulized SUN-101 using an Investigational eFlow® Closed System (CS) nebulizer in subjects with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD 2014) guidelines.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter, efficacy and safety trial of 12 weeks of treatment with nebulized SUN-101 using an Investigational eFlow® Closed System (CS) nebulizer in approximately 645 subjects with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD 2014) guidelines.

SUN-101 or placebo will be administered twice daily as an oral inhalation using the investigational eFlow CS nebulizer. Approximately 150 subjects will be enrolled in the substudy (at selected sites only). These subjects will be required to participate in serial spirometry, vital signs, ECGs, and an additional Holter monitor assessment at Visit 6 (Week 12). This subset of subjects will be referred to as the Substudy Population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 40 years, inclusive
2. A clinical diagnosis of COPD according to the GOLD 2014 guidelines
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, or equivalent)
4. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1 < 80% of predicted normal and > 0.7 L during Screening (Visit 1)
5. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio < 0.70 during Screening (Visit 1)
6. Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines (2005)
7. Subject, if female ≤ 65 years of age and of child bearing potential, must have a negative serum pregnancy test at Visit 1. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a) an oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following participation; b) barrier method of contraception, eg, condom and /or diaphragm with spermicide while participating in the study; and/or c) abstinence
8. Willing and able to provide written informed consent
9. Willing and able to attend all study visits and adhere to all study assessments and procedures

Exclusion Criteria:

1. Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject
2. Concomitant clinically significant respiratory disease other than COPD (eg, asthma, tuberculosis, bronchiectasis or other non-specific pulmonary disease).
3. Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to Screening (Visit 1)
4. Use of daily oxygen therapy > 12 hours per day
5. Respiratory tract infection within 6 weeks prior to Screening (Visit 1)
6. Use of oral, intravenous, or intramuscular steroids within 3 months prior to Screening (Visit 1)
7. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin
8. Prolonged QTcF (> 450 msec for males and > 470 msec for females) during Screening (Visit 1) as determined from the report provided by the central laboratory, or history of long QT syndrome
9. History of or clinically significant ongoing bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months.
10. History of narrow angle glaucoma
11. History of hypersensitivity or intolerance to aerosol medications
12. Recent documented history (within the previous 3 months) of substance abuse
13. Significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator
14. Participation in another investigational drug study where drug was received within 30 days prior to Screening (Visit 1) or current participation in another investigational drug trial, including a SUN-101 study
15. Previously received SUN-101 (active treatment; formerly known as EP-101).
16. Contraindicated for treatment with, or having a history of reactions/hypersensitivity to anticholinergic agents, beta2 agonists, or sympathomimetic amines

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sunovion Respiratory Director
Locations (44):
- United States (44):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Clinical Research Consortium - Arizona, Tempe, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Clermont Medical Research, Clermont, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research, Kissimmee, Florida
  - AppleMed Research, Inc., Miami, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Emerald Coast Research Associates, Panama City, Florida
  - Clinical Research of West Florida, Inc, Tampa, Florida
  - Abraham Reasearch, PLLC, Fort Mitchell, Kentucky
  - Pulmonary Research Institute of Southeast Michigan, Livonia, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - Midwest Chest Consultants, P.C., Saint Charles, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - AAIR Research Center, Rochester, New York
  - American Health Research, Inc., Charlotte, North Carolina
  - Hickory Research Center, Hickory, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Columbus Regional Research Institute, Columbus, Ohio
  - Columbus Clinical Research, Inc, Columbus, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Palmetto Medical Research Associates, LLC, Easley, South Carolina
  - Greenville Pharmaceutical Research, Inc, Greenville, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Piedmont Research Partners, LLC, Old Point Station, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - CU Pharmaceutical Research, Union, South Carolina
  - Texas Pulmonary and Critical Care Consultants, PA, Fort Worth, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Pulmonary Research of Abingdon, LLC, Abingdon, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia

REFERENCES:
- [Result] Kerwin E, Donohue JF, Goodin T, Tosiello R, Wheeler A, Ferguson GT. Efficacy and safety of glycopyrrolate/eFlow(R) CS (nebulized glycopyrrolate) in moderate-to-very-severe COPD: Results from the glycopyrrolate for obstructive lung disease via electronic nebulizer (GOLDEN) 3 and 4 randomized controlled trials. Respir Med. 2017 Nov;132:238-250. doi: 10.1016/j.rmed.2017.07.011. Epub 2017 Jul 19. PMID 28838685
- [Derived] Ohar J, Tosiello R, Goodin T, Sanjar S. Efficacy and safety of a novel, nebulized glycopyrrolate for the treatment of COPD: effect of baseline disease severity and age; pooled analysis of GOLDEN 3 and GOLDEN 4. Int J Chron Obstruct Pulmon Dis. 2018 Dec 18;14:27-37. doi: 10.2147/COPD.S184808. eCollection 2019. PMID 30587959
- [Derived] Ferguson GT, Kerwin EM, Donohue JF, Ganapathy V, Tosiello RL, Bollu VK, Rajagopalan K. Health-Related Quality of Life Improvements in Moderate to Very Severe Chronic Obstructive Pulmonary Disease Patients on Nebulized Glycopyrrolate: Evidence from the GOLDEN Studies. Chronic Obstr Pulm Dis. 2018 Jun 6;5(3):193-207. doi: 10.15326/jcopdf.5.3.2017.0178. PMID 30584583

RESULTS

PARTICIPANT FLOW:
Period: All Collected
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Started | 218 | 217 | 218
Completed | 201 | 203 | 191
Not Completed | 17 | 14 | 27
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 3
Not completed — Withdrawal by Subject | 11 | 11 | 22
Not completed — invetigator disretion | 2 | 0 | 0
Not completed — instillation site pain | 0 | 0 | 1
Not completed — exacerbation of COPD | 0 | 0 | 1
Not completed — moved/travel | 0 | 1 | 0
Period: On Study Treatment
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Started | 218 | 217 | 218
Completed | 191 | 194 | 176
Not Completed | 27 | 23 | 42
Not completed — Lack of Efficacy | 2 | 3 | 4
Not completed — non-compliance with study medication | 0 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 3 | 5
Not completed — move/travel | 2 | 6 | 5
Not completed — dissastisfaction with device | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — investigator discretion | 2 | 0 | 0
Not completed — durg not working | 0 | 1 | 1
Not completed — Adverse Event | 10 | 8 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer | Total
Number analyzed (Participants) | 218 | 217 | 218 | 653
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 135 | 122 | 109 | 366
  >=65 years | 83 | 95 | 109 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.09) | 63.1 (8.78) | 63.7 (8.37) | 63.1 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 99 | 107 | 304
  Male | 120 | 118 | 111 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 6 | 19
  Not Hispanic or Latino | 212 | 210 | 212 | 634
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 18 | 15 | 20 | 53
  White | 198 | 200 | 196 | 594
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 218 | 217 | 218 | 653
cardiovascular risk (low/high) and categories for high caridovascular risk [Count of Participants; unit: Participants] — Cardiovascular risk was stratified as low versus high risk where the high risk stratum was defined as any participant with a pre-existing diagnosis of ischemic heart cardiovascular risk disease, cerebrovascular disease, peripheral arterial disease, hypertension, clinically significant arrhythmia or heart failure.
  Participants
    low cardiovascular risk | 77 | 78 | 76 | 231
    high cardiovascular risk | 141 | 139 | 142 | 422
    cerebrovascular disease | 10 | 13 | 14 | 37
    peripheral arterial disease | 10 | 13 | 14 | 37
    clinically significant arrhythmia | 7 | 13 | 2 | 22
    heart failure | 9 | 7 | 8 | 24
    hyertension | 127 | 128 | 138 | 393
background long-acting beta(2) agonist (LABA) use [Count of Participants; unit: Participants] — background LABA [+/- ICS] use was stratified as "yes" or "no" where the continuation of background therapy, in approximately 30% of the study population, required the subject to be on a stable dose of the medication for 4 weeks prior to study entry.
  Participants
    background LABA use =yes | 68 | 66 | 63 | 197
    background LABA use =no | 150 | 151 | 155 | 456
Forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: liters] — spirometry was performed according to internationally accepted standards. Baseline FEV1 is defined as the mean of the two dose values at 45 and 15 minutes prior to first dose.
  liters | 1.3745 (0.52957) | 1.3108 (0.50243) | 1.3122 (0.47511) | 1.3325 (0.50297)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: ALL COLLECTED-Spirometry was performed according to internationally accepted standards.Trough FEV1 at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.Change from baseline in trough FEV1 was calculated as the trough FEV1 value at Week 12 minus the morning trough FEV1 at baseline (mean of the two pre-dose values at 45 and 15 minutes prior to the first dose). All collected values were used in this analyses, regardless if the subject remained on randomized treatment or not, and regardless if the values might potentially be affected by other therapies or not Values not collected remained as missing values and were assumed to be missing at random (MAR) "ALL COLLECTED" and "ON TREATMENT" data are the same. The only difference is in the number of visits included for those participants who may have discontinued randomized treatment but remained in the study." for all endpoints
Time Frame: Baseline and Week 12
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study medication. Subjects were analyzed based on the treatment they were randomized to.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
liters | 0.0961 (0.01371) | 0.0886 (0.01369) | -0.0075 (0.01397)
Statistical Analysis 1: Comparison: SUN-101 50 mcg BID eFlow (CS) Nebulizer vs Placebo BID eFlow (CS) Nebulizer; The change from baseline in trough FEV1 was analyzed using a mixed model for repeated measures including terms for treatment, cardiovascular risk, background LABA use, visit, visit by treatment interaction, and baseline FEV1 as a covariate. An unstructured covariance matrix was used; Test type: Superiority — A sample size of 215 subjects per treatment would give ~ 90% power to detect a treatment difference of 80 mL in the change from baseline in trough FEV1 at Week 12 between each of the 2 SUN-101 dose groups and placebo at alpha= 0.05, assuming a standard deviation of 255 mL and using a 2-sided test; p < 0.0001, MMixed Model Repeat Measurement — The primary null hypothesis for this study is that the mean change from baseline in trough FEV1 at Week 12 for the SUN-101 50 mcg dose is equal to the mean change from baseline in trough FEV1 at Week 12 for Placebo; to control the family-wise Type I error rate,the Hochberg procedure(a tree-structured gatekeeping procedure)was used for comparisons of this endpoint; Least Squares Mea Difference (SE) = 0.1036, 95% CI 2-sided [0.0663 to 0.1409], Standard Error of Mean 0.01900 — standard error of the least squares mean
Statistical Analysis 2: Comparison: SUN-101 25 mcg BID eFlow (CS) Nebulizer vs Placebo BID eFlow (CS) Nebulizer; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; to control the family-wise Type I error rate,the Hochberg procedure(a tree-structured gatekeeping procedure)was used for comparisons of the endpoint; Least Squares Mean Difference (SE) = 0.0961, 95% CI 2-sided [0.0589 to 0.1334], Standard Error of Mean 0.01896 — Standard error of the least squares mean

2. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) Week 12
Description: ON TEATMENT-Spirometry was performed according to internationally accepted standards.Trough FEV1 at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.Change from baseline in trough FEV1 was calculated as the trough FEV1 value at Week 12 minus the morning trough FEV1 at baseline (mean of the two pre-dose values at 45 and 15 minutes prior to the first dose).Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
liters | 0.1025 (0.01497) | 0.0814 (0.01475) | -0.0238 (0.01534)
Statistical Analysis 1: Comparison: SUN-101 50 mcg BID eFlow (CS) Nebulizer vs Placebo BID eFlow (CS) Nebulizer; The change from baseline in trough FEV1 was analyzed using mixed model repeated measures including terms for treatment, cardiovascular risk, background LABA use, visit week, visit week by treatment interaction, and baseline FEV1 as a covariate. An unstructured covariance matrix was used; Test type: Superiority; p < 0.0001, Least squares mean (SE) — In order to control the family-wise Type I error rate, the Hochberg procedure (a tree-structured gatekeeping procedure) was used for comparisons of the primary efficacy endpoints and the key secondary efficacy endpoints; Least Squares Mean (SE) = 0.1264, 95% CI 2-sided [0.0856 to 0.1672], Standard Error of Mean 0.02076
Statistical Analysis 2: Comparison: SUN-101 25 mcg BID eFlow (CS) Nebulizer vs Placebo BID eFlow (CS) Nebulizer; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — In order to control the family-wise Type I error rate, the Hochberg procedure (a tree-structured gatekeeping procedure) was used for comparisons of the primary efficacy endpoints and the key secondary efficacy endpoints; p < 0.0001, LS mean (SE); LS mean (SE) = 0.1052, 95% CI 2-sided [0.0647 to 0.1457], Standard Error of Mean 0.02060

3. Secondary Outcome: Standardized Change From Baseline at Week 12 in FEV1 Area Under the Curve (AUC) (0-12) in the Substudy Population
Description: ALL COLLECTED The standardized FEV1 AUC(0-12) was calculated at weeks 0 and 12 for the Substudy Population with extended spirometry measurements. The trapezoidal rule was used to calculate FEV1 AUC and then normalized to the length of time. Intermittent missing spirometry measurements were ignored and the trapezoidal rule would simply span the missing time point(s). If the Hour 12 time point was missing, then the AUC(0-12) calculation was based on the time interval up to the last non-missing time point prior to Hour 12. If a subject has a missing baseline FEV1, then that subject had a missing AUC. All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not, and regardless if the values might potentially be affected by other therapies or not Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: The Substudy Population consisted of all ITT subjects who participated in post-dose serial measurements
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 62 | 49 | 42
liters | 0.0749 (0.02638) | 0.0579 (0.3011) | -0.0474 (0.03229)

4. Secondary Outcome: Standardized Change From Baseline at Week 12 in FEV1 Area Under the Curve (AUC) (0-12) in Substudy Population
Description: ON TREATMENT The standardized FEV1 AUC(0-12) was calculated at weeks 0 and 12 for the Substudy Population with extended spirometry measurements. The trapezoidal rule was used to calculate FEV1 AUC and then normalized to the length of time. Intermittent missing spirometry measurements were ignored and the trapezoidal rule would simply span the missing time points. If the Hour 12 time point was missing, then the AUC(0-12) calculation was based on the time interval up to the last non-missing time point prior to Hour 12. If a subject has a missing baseline FEV1, then that subject had a missing AUC.Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: The Substudy Population consisted of all ITT subjects who participated in post-dose serial measurements, including serial spirometry, serial ECGs, serial vital sign measurements, as well as Holter monitoring at Visit 6.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 62 | 49 | 42
liters | 0.0708 (0.02792) | 0.0496 (0.03280) | -0.0527 (0.03450)

5. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Week 12
Description: ALL COLLECTED Spirometry was performed according to internationally accepted standards. Trough FVC at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not, and regardless if the values might potentially be affected by other therapies or not Values not collected remained as missing values and were assumed to be missing at random
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
liters | 0.1476 (0.02226) | 0.1515 (0.02220) | 0.0147 (0.2266)

6. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) Week 12
Description: ON TREATMENT Spirometry was performed according to internationally accepted standards. Trough FVC at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose. Change from baseline in trough FVC was calculated as the trough FVC value at Week 12 minus the morning trough FVC at baseline (mean of the two pre-dose values at 45 and 15 minutes prior to the first dose).Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
liters | 0.1566 (0.02392) | 0.1393 (0.02353) | -0.0101 (0.2450)

7. Secondary Outcome: Change From Baseline in Health Status Measured by St. George's Respiratory Questionnaire (SGRQ) at Week 12/End of Study
Description: ALL COLLECTED Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: symptoms, activity, and impacts. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is 0 and the highest 100. Higher values correspond to greater impairment of health status.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
scores on a scale | -2.363 (0.8344) | -4.250 (0.8211) | -0.844 (0.8396)

8. Secondary Outcome: Change From Baseline in Health Status Measured by St. George's Respiratory Questionnaire (SGRQ) Week 12/End of Study
Description: ON TREATMENT Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: symptoms, activity, and impacts. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is 0 and the highest 100. Higher values correspond to greater impairment of health status.
  Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
scores on a scale | -2.538 (0.8391) | -3.762 (0.8187) | -0.690 (0.8535)

9. Secondary Outcome: Change in Number of Rescue Medication Puffs Per Day Over the 12-week Double-blind Treatment Period
Description: ALL COLLECTED Participants completed an electronic diary (eDiary) daily (night time) to record the number of puffs of rescue medication inhaled in the previous 24 hours. A negative change from baseline indicates improvement.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Week 0-12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: puffs (medication used)
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
puffs (medication used) | -0.815 (0.1234) | -0.609 (0.1259) | -0.632 (0.1257)

10. Secondary Outcome: Number of Subjects With Major Adverse Cardiac Events (MACE)
Description: ALL COLLECTED All deaths and any other findings suggestive of a potential MACE (including clinically relevant information and SAEs, and all PTs form the SMQs "myocardial infarction", "other ischemic heart disease", "central nervous system hemorrhages and cerebrovascular conditions") were sent to an adjudication committee for review and categorized as CV death, nonfatal MI, and nonfatal stroke. The MACE score was defined as the total number of subjects with CV deaths, nonfatal MIs, and nonfatal strokes. These events were collected for the double-blind period (from the first date of study medication until the date of last contact)
Time Frame: Week 0-12
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
participants
  MACE score | 3 | 0 | 0
  Cardiovascular Death | 1 | 0 | 0
  non-fatal myocardial infraction | 1 | 0 | 0
  non-fatal stroke | 1 | 0 | 0

11. Secondary Outcome: Percentage of Subjects With Major Cardiac Events (MACE)
Description: as for outcome 10
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
percentage of participants
  MACE score | 1.4 | 0 | 0
  Cardiovascular Death | 0.5 | 0 | 0
  non-fatal myocardial infraction | 0.5 | 0 | 0
  non-fatal stroke | 0.5 | 0 | 0

12. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: ON TREATMENT A TEAE is defined as any non-serious AE that occurred on or after the first dose of study medication and within 7 days after the last dose of study medication, or any serious AE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent AE is an on-treatment AE.
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
participants | 105 | 86 | 114

13. Secondary Outcome: Percent of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: as for outcome 12
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
percentage of participants | 48.2 | 39.6 | 52.3

14. Secondary Outcome: Number of Subjects With Treatment Emergent Serious Adverse Events (SAE)
Description: ON TREATMENT A treatment emergent SAE is defined as any SAE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent SAE is an on-treatment SAE
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
participants | 10 | 8 | 11

15. Secondary Outcome: Percent of Subjects With Treatment Emergent Serious Adverse Events (SAE)
Description: as for outcome 14
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
percentage of participants | 4.6 | 3.7 | 5.0

16. Secondary Outcome: Number of Subjects Who Discontinue Treatment Due to TEAE
Description: ON TREATMENT A TEAE is defined as any AE that occurred on or after the first dose of study medication and within 7 days after the last dose of study medication, or any serious AE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent AE is an on-treatment AE.
Time Frame: Week 0-12
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study meidcation
Measure: Number; unit: participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
participants | 8 | 7 | 21

17. Secondary Outcome: Percent of Subjects Who Discontinue Treatment Due to TEAE
Description: as for outcome 16
Time Frame: Week 0-12
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
percentage of participants | 3.7 | 3.2 | 9.6

18. Secondary Outcome: Incidence Rate Per 100 Person-years of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: ALL COLLECTED All deaths and any other findings suggestive of a potential MACE (including clinically relevant information and SAEs, and all PTs form the SMQs "myocardial infarction", "other ischemic heart disease", "central nervous system hemorrhages and cerebrovascular conditions") were sent to an adjudication committee for review and categorized as CV death, nonfatal MI, and nonfatal stroke. The MACE score was defined as the total number of subjects with CV deaths, nonfatal MIs, and nonfatal strokes. These events were collected for the double-blind period (from the first date of study medication until the date of last contact)I ncidence rate: TT= Total Time in years. Total Time (TT) is defined as the time from the first date of study drug until the latter of the date of last contact or 30 days after the date of last dose. Incidence Rate (per 1000 person-years) = n/TT x 1000.
Time Frame: Week 0-12
Population: as for outcome 10
Measure: Number; unit: events per 100 person-years
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Number analyzed (Participants) | 218 | 217 | 218
events per 100 person-years
  MACE score | 45.5 | 0 | 0
  Cardiovascular Death | 15.2 | 0 | 0
  non-fatal myocardial infraction | 15.2 | 0 | 0
  non-fatal stroke | 15.2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0-12
Description: A treatment emergent SAE is defined as any SAE that occurred on or after the first dose of study medication and within 30 days after the last does of study medication. A treatment emergent SAE is an on-treatment SAE
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID eFlow (CS) Nebulizer | Placebo BID eFlow (CS) Nebulizer
Serious Adverse Events (participants affected / at risk) | 10/218 | 8/217 | 11/218
Other Adverse Events (participants affected / at risk) | 37/218 | 23/217 | 38/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=218) | SUN-101 25 mcg BID eFlow (CS) Nebulizer (N=217) | Placebo BID eFlow (CS) Nebulizer (N=218)
angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
gallbladder necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
lobar pheumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
antiphospholiid antibodies (Investigations) | 0 (0) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
malignant neoplasm of pleura metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=218) | SUN-101 25 mcg BID eFlow (CS) Nebulizer (N=217) | Placebo BID eFlow (CS) Nebulizer (N=218)
chronic obstructive ulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 9 (9) | 17 (19)
cough (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 16 (20) | 22 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.